CLINICAL TRIAL: NCT05981924
Title: Effects of Music Therapy on Perioperative Anxiety and Pain Management in Lung Surgery: A Randomized, Prospective, Multidisciplinary Trial
Brief Title: Perioperative Music Therapy Plus Oxycodone in Perioperative Management of Lung Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hao Long (Other)
Collaborators: Sun Yat-sen University School of Art (Unknown); Sun Yat-sen University Department of Psychology (Unknown)
Responsible Party: Sponsor-Investigator, Hao Long, Prof., Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A2023-003
Record Dates: First submitted 2023-07-31; First posted 2023-08-08 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Analgesia; Lung Cancer
Keywords: Music Therapy; Anxiety; Quality of Life
MeSH Terms: conditions — Agnosia; Lung Neoplasms; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned into two groups, the experimental group will receive music therapy and oxycodone for the pain management after thoracic surgery. The control group will only use oxycodone to relief the pain.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxycodone with Perioperative Music Therapy (Experimental): Using perioperative music therapy plus oxycodone to manage the postoperative pain
  Interventions: Other: Perioperative Music Therapy
- Oxycodone without Perioperative Music Therapy (No Intervention): Using oxycodone only to manage the postoperative pain

INTERVENTIONS:
Other: Perioperative Music Therapy — Music therapist will play customized music in the perioperative period on the basis of oxycodone analgesia
  Arms: Oxycodone with Perioperative Music Therapy

SUMMARY:
To explore the feasibility and effectiveness of Perioperative Music Therapy Plus Oxycodone in pain management after thoracic surgery, patients will be randomly assigned into two groups. The experimental group will receive perioperative music therapy and the control group will not. We will record and contrast the postoperative oxycodone usage to evaluate the effect of music therapy in relieving the pain. We will also use visual analogue scale, questionnaire and EEG to evaluate patients' anxiety and depression.

ELIGIBILITY:
Inclusion Criteria:

* Enhanced CT or PET/CT indicate primary malignant pulmonary nodule;
* The clinical stage belongs to cT1-4N0-2M0 before treatment or ycT1-4N0-2M0 after neoadjuvant treatment (AJCC/TNM 8th Edition);
* Suitable for video-assisted thoracoscopic surgery after evaluated by thoracic surgeon;
* FEV1 > 1.5L and DLCO > 60% pred;
* Hearing loss lesser than 35 decibels (dB) in the better hearing ear;
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2;
* American Society of Anesthesiologists Score of 1 or 2;
* Confirmed eligibility for R0 resection for curative intent by thoracic surgeon assessment;
* Adequate cardiopulmonary function, confirmed to meet the requirement for surgical resection for curative intent;
* Able to provide written informed consent and able to understand and agree to comply with study requirements and evaluation forms;
* Life expectancy greater than 12 months

Exclusion Criteria:

* Enhanced CT or PET/CT indicate metastatic malignant pulmonary nodule;
* Hearing loss greater than 35 decibels (dB) in the better hearing ear;
* Active autoimmune disease or history of autoimmune disease that may recur; Note: well-controlled type 1 diabetes is allowed; hypothyroidism (controlled with thyroid hormone replacement only); well-controlled celiac disease; skin disease not requiring systemic treatment (eg, vitiligo, psoriasis, alopecia); any other condition that is not expected to recur in the absence of an external trigger.
* History of interstitial lung disease, pneumonitis or uncontrolled systemic diseases, including diabetes, hypertension, pulmonary fibrosis, acute lung disease;
* Serious infection occurred before grouping, including but not limited to hospitalization due to infectious complications, bacteremia or severe pneumonia; severe chronic or active infection (including pulmonary tuberculosis infection, etc.) requiring systemic (oral or intravenous) antibiotics within 14 days before grouping;
* Simultaneous participation in another therapeutic clinical study;
* Pregnant or lactating women, or male and female patients planning to have children during the study;
* Other conditions that the investigators consider inappropriate for participation in this trial, such as poor compliance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-04-20 (Actual)

PRIMARY OUTCOMES:
The total dose of oxycodone within 48 hours after surgery | 48 hours after surgery
  The total dose of oxycodone within 48 hours after surgery

SECONDARY OUTCOMES:
The VSA-A Score | From 1 day before surgery to the third day after surgery
  The Visual Analogue Scale-Anxiety Score at different observation point
The VSA-P Score | From the first day to the third day after surgery
  The Visual Analogue Scale-Pain Score at different observation point
The incidence rate of analgesic related adverse reaction | 48 hours after surgery
  The incidence rate of analgesic related adverse reaction within 72 hours after surgery
The usage of extra analgesics after surgery | 48 hours after surgery
  The usage of extra analgesics after surgery, such as Parecoxib, Tramadol or Morphine
The kind and usage of anesthetics for anesthesia induction and maintenance | During the surgery
  The kind and usage of anesthetics for anesthesia induction and maintenance, such as Propofol, Sufentanil and Cisatracurium
The quality of life after treatment | The third day after surgery
  The quality of life assessed by questionnaire on the third day after surgery
The press times of PCIA pump within 48 hours after surgery | 48 hours after surgery
  The press times of PCIA pump within 48 hours after surgery

OTHER OUTCOMES:
Changes of resting beta power of electroencephalography in the central brain areas by preoperative treatment | 1 hour before surgery
  Changes of resting beta power of electroencephalography in the central brain areas by preoperative treatment
Changes of resting beta power of electroencephalography in the frontal midline brain areas by preoperative treatment | 1 hour before surgery
  Changes of resting beta power of electroencephalography in the frontal midline brain areas by preoperative treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Palmer JB, Lane D, Mayo D, Schluchter M, Leeming R. Effects of Music Therapy on Anesthesia Requirements and Anxiety in Women Undergoing Ambulatory Breast Surgery for Cancer Diagnosis and Treatment: A Randomized Controlled Trial. J Clin Oncol. 2015 Oct 1;33(28):3162-8. doi: 10.1200/JCO.2014.59.6049. Epub 2015 Aug 17. PMID 26282640
- [Result] Zhou W, Ye C, Wang H, Mao Y, Zhang W, Liu A, Yang CL, Li T, Hayashi L, Zhao W, Chen L, Liu Y, Tao W, Zhang Z. Sound induces analgesia through corticothalamic circuits. Science. 2022 Jul 8;377(6602):198-204. doi: 10.1126/science.abn4663. Epub 2022 Jul 7. PMID 35857536